CLINICAL TRIAL: NCT07234565
Title: The Effects of "Social Optimization Chat for Interactive Learning for Heart Failure" (SOCIAL_HF) on Improving Social Frailty: A Randomized Controlled Trial
Brief Title: SOCIAL_HF: Improving Social Frailty Through Interactive Learning
Acronym: SOCIAL_HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 25-387
Record Dates: First submitted 2025-09-21; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Social frailty; Heart Failure; WeChat-based; Interactive learning; Self-care; Social support; Social participation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): One educational booklet
  Interventions: Other: Self-study heart failure self-care manual
- SOCIAL_HF (Experimental): One educational booklet; one session per week, each lasting one hour, with two sessions in the final week, totaling seven online group sessions; daily 0.5-hour WeChat group chats, five days a week.
  Interventions: Behavioral: SOCIAL_HF

INTERVENTIONS:
Behavioral: SOCIAL_HF — Participants will engage in a 6-week, WeChat-based group learning program called SOCIAL_HF, focused on heart failure self-care. This program comprises two key components: structured real-time interactive learning and ongoing synchronous support. Real-time interactive learning will be conducted through WeChat video group meetings weekly, featuring peer sharing, problem-solving collaborative tasks, health goal setting, progress sharing, and the establishment of group contracts. Daily synchronous chat interactions will revolve around completing group contract tasks, weekly quizzes, and daily sharing. Additionally, participants will have access to an online self-care resource hub on the WeChat platform for reference and use.
  Arms: SOCIAL_HF
Other: Self-study heart failure self-care manual — The control group will establish a WeChat connection with PI and receive standard care, which includes a health education manual. However, they will not participate in group learning or discussions. They can consult with research assistants via WeChat for any questions they may have, but the researchers will only provide explanations related to the health education manual and will not offer additional educational resources or group interactions.
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to learn whether the WeChat-based program "Social Optimization Chat for Interactive Learning for Heart Failure" (SOCIAL_HF) can improve social frailty in elderly patients with heart failure. The main questions it aims to answer are:

Can a 6-week WeChat online group interactive learning program (SOCIAL_HF) improve social frailty? Does the intervention enhance self-care abilities, social participation, and perceived social support? Researchers will compare SOCIAL_HF to usual care (self-study heart failure self-care manual) to assess whether SOCIAL_HF can improve social functioning.

Participants will:

Engage in weekly WeChat video meetings for six weeks (Participate in peer sharing and collaborative tasks).

Complete daily health task check-ins. Access online self-care resources.

DETAILED DESCRIPTION:
Background: Patients with heart failure often face challenges such as shortness of breath, fatigue, and decline in daily functioning, significantly affecting their social activities and resource access, leading to social frailty. Research indicates that social frailty not only lowers quality of life but may also negatively impact survival outcomes. However, effective interventions addressing this issue remain scarce.

Aims: This study aims to improve social frailty among heart failure patients by enhancing social resources and promoting social activities. The specific objective is to evaluate the effectiveness of a 6-week WeChat online group interactive learning program (SOCIAL_HF), which is designed to increase participant interaction and social networks, thereby improving self-care abilities and breaking the vicious cycle of social frailty.

Methods: This study will be a two-arm, single-blind, randomized controlled trial (RCT), with a planned recruitment of 208 participants. The study comprises two phases: a feasibility study and a larger-scale RCT. Both phases will use the same recruitment and intervention procedures, with the main differences being the timepoints of follow-ups. Recruitment will occur through face-to-face interviews at multiple hospitals in Shanghai, with eligible participants randomly assigned to either the control group (usual care) or the 6-week intervention group in a 1:1 ratio. The random sequence will be generated by an independent research assistant using a computer-based randomization program. The generated numbers will be placed in opaque envelopes and allocated sequentially by the PI on-site. The intervention will include weekly WeChat video meetings, peer sharing, collaborative tasks, and health goal reviews, as well as daily health task check-ins and access to online self-care resources. The control group will establish a WeChat connection with the research assistants and receive standard care, which includes a health education manual. However, they will not participate in group learning or discussions.

During the feasibility study phase, participants will undergo primary and secondary outcome assessments at baseline and immediately post-intervention, conducted by independent research assistants. A mixed-methods approach will be employed to assess feasibility, including quantitative and qualitative analyses to evaluate recruitment status, attendance, and retention rates. Additionally, one-on-one semi-structured interviews will be conducted to determine the appropriateness and acceptability of the intervention measures. In the large-scale RCT phase, participants will receive outcome assessments at baseline, immediately post-intervention, and three months after the intervention to evaluate its maintenance effects on primary and secondary outcomes.

Outcomes: The primary outcome is social frailty, and the secondary outcome is perceived social support, social participation, and self-care.

ELIGIBILITY:
Inclusion Criteria:

1. 60 years old and above;
2. Live in the community;
3. a definitive diagnosis of heart failure based on the Framingham Heart Failure Diagnostic Criteria;
4. a diagnosis of heart failure for 6 months or longer;
5. evidence of social pre-frailty or frailty, determined by the SFS-8 score ≥ 2; (6) possession of a smartphone and experience using WeChat;

(7) be able to read and write Chinese.

Exclusion Criteria:

1. severe cognitive impairment or dementia;
2. known mental illnesses;
3. any communication barriers may hinder participation in SOCIAL_HF, such as illiteracy, reading disabilities, speak local dialect only, and difficulties in language comprehension;
4. any sensory impairments that may affect learning or interaction with others on WeChat, including untreated severe hearing loss and vision impairments；
5. are currently participating in other intervention studies.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Social frailty | Feasibility study phase: At enrollment and immediately post-intervention. During full RCT phase: At enrollment, immediately post-intervention and 3-month post-intervention.
  Social frailty will be assessed by using Social Frailty Scale-8 item developed by Pek in Singapore. It consists of eight questions covering whether they visit friends sometimes, seek advice from family and friends, have people they can trust, go out less frequently, eat alone, have financial difficulties, live alone, talk to someone every day. It uses a dichotomous scoring method with a total score ranging from 0 to 8 points. A score of 0-1 indicates social non-frailty (SNF), 2-3 indicates social pre-frailty (SPF), and ≥4 indicates social frailty (SF).

SECONDARY OUTCOMES:
Perceived social support | Feasibility study phase: At enrollment and immediately post-intervention. During full RCT phase: At enrollment, immediately post-intervention and 3-month post-intervention.
  Perceived social support as an indicator of social resources will be assessed by the Chinese Mandarin version of the Medical Outcomes Study Social Support Survey (MOS-SSS-CM), which consists of 19 items across four dimensions: tangible support (4 items), informational and emotional support (8 items), positive social interaction (4 items), and affectionate support (3 items). Each item is rated on a 5-point Likert scale, with higher scores indicating better support.
Social participation | Feasibility study phase: At enrollment and immediately post-intervention. During full RCT phase: At enrollment, immediately post-intervention and 3-month post-intervention.
  Social participation serves as an indicator of engagement in social activities. The Impact on Participation and Autonomy Questionnaire (IPA), which is a self-report instrument that measures people's perceptions of participation and autonomy, will be used to evaluate the social participation of older adults with heart failure. The original scale has a Cronbach's α ranging from 0.81 to 0.9. The Chinese version of the questionnaire was translated by Li et al [48]. Comprising 25 items, the scale is organized into four distinct dimensions: autonomy indoors (7 items), family role (7 items), autonomy outdoors (5 items), and social life (6 items). A 5-point Likert scale is utilized, with "a lot" receiving 0 points and "a little" receiving 4 points. Scores can range from 0 to 100, where a higher score reflects a lower level of social participation.
Self-care | Feasibility study phase: At enrollment and immediately post-intervention. During full RCT phase: At enrollment, immediately post-intervention and 3-month post-intervention.
  Self-care will be assessed by the Chinese version of the Self-care Heart Failure Index version 7.2 (SCHFI v7.2-C), which comprises 29 items across three dimensions. Scores range from 0 to 100, with 70 or above indicating adequate self-care.

OTHER OUTCOMES:
Feasibility indicators | Recruitment Status: Assessed at baseline. Attendance Rate: Monitored during the intervention phase (from enrollment through the 6-week intervention period). Retention Rate: Through study completion, an average of 6 months.
  For the feasibility study, research team will comprehensively assess the feasibility through recruitment status, attendance, and retention rates.
Appropriateness, practicality, and acceptability of the intervention measures | Within two weeks after completion of the intervention
  One-on-one semi-structured interviews will be conducted to evaluate the appropriateness, practicality, and acceptability of the intervention measures. The interviews will focus on three areas: (1) Appropriateness: Assessing whether the intervention meets participants' needs and expectations; (2) Practicality: Evaluating the feasibility of the intervention in real-world settings, including participants' experiences; (3) Acceptability: Understanding participants' overall perceptions, including satisfaction, engagement factors, and potential barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Miao Miao, MN, RN, Principal Investigator — School of Nursing, University of Hong Kong
Locations (3):
- China (3):
  - Fudan University Affiliated Huadong Hospital, Shanghai
  - Shanghai Baoshan District Integrated Traditional Chinese and Western Medicine Hospital, Shanghai
  - Shanghai Jiao Tong University School of Medicine Affiliated Songjiang Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
We will share the following specific individual participant data (IPD): age, gender, residential status, marital status, medical history, and targeted outcomes.
Supporting Information: Study Protocol
Time Frame: The individual participant data (IPD) that underlie the results reported in this article will be made available upon acceptance of the manuscript for publication. The data will be accessible for a minimum of 5 years from the date of publication.
Access Criteria: The de-identified IPD will be available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Access requests will be reviewed by a designated data access committee (or by the corresponding author) to ensure the proposed use is scientifically valid and does not conflict with the original informed consent.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT07234565/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT07234565/ICF_001.pdf